CLINICAL TRIAL: NCT03645941
Title: Social Media Intervention to Promote Smoking Treatment Utilization and Cessation Among Alaska Native Smokers
Brief Title: Connecting Alaska Native People to Quit Smoking
Acronym: CAN Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-009947; R34DA046008 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-24 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Smoking Cessation; Smoking, Cigarette; Smoking, Tobacco; Smoking
Keywords: Social Media; Alaska Native
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Smoking Cessation; Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: Our approach follows the three-stage model of behavioral therapies development and the proposed aims correspond to the two sub-stages characterizing Stage I work. In Stage Ia formative work, we will develop the Facebook intervention. In Stage Ib, we will use rigorous design and methodology to evaluate the intervention's feasibility and potential efficacy. Stage Ib results will inform a future R01, Stage II, randomized efficacy trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quitline/Treatment Referral (No Intervention): Description of tobacco treatment services, phone numbers and web links sent via postal mail (printed materials) and email. Treatment options provide free, professional assistance based on U.S. clinical practice guidelines: (1)AK quitline, (2)regional tribal tobacco cessation programs, and (3)smokefree.gov resources (e.g., free texting program and smartphone application, quit guide)
- Facebook+Quitline/Treatment Referral (Experimental): * Participants join a secret/private, culturally relevant Facebook group moderated by an AN tobacco research counselor for 3 months
  * Once daily moderator postings for 30 days, repeated each month for 3 months; plus 3-4 daily check-ins/postings to respond to participant generated content and encourage sharing of personal stories/experiences relevant to all stages of the quitting process and treatment engagement
  * Description of tobacco treatment services, phone numbers and web links sent via postal mail (printed materials) and email. Treatment options provide free, professional assistance based on U.S. clinical practice guidelines: (1)AK quitline, (2)regional tribal tobacco cessation programs, and (3)smokefree.gov resources (e.g., free texting program and smartphone application, quit guide)
  Interventions: Behavioral: Facebook Group

INTERVENTIONS:
Behavioral: Facebook Group — The pilot trial, a two-arm, parallel groups, randomized controlled design, will enroll 60 participants randomized with 1:1 allocation to the intervention or control condition. Participants will be randomized within stratified blocks based on sex (male, female), age group (19-29, 30-49, 50+ years), and region (urban, rural); potential variables related to outcomes. Assessments will be conducted for both study groups at baseline and at 1, 3, and 6 month follow-up.
  Arms: Facebook+Quitline/Treatment Referral

SUMMARY:
The prevalence of smoking among US adults is highest among American Indians and Alaska Native (AI/AN) persons; however, there are a lack of tobacco cessation interventions developed specific to this disparity group. Social media holds promise as a scalable intervention strategy to promote engagement in treatment and cessation outcomes for Alaska Native (AN) people.

Researchers plan to develop and pilot test a culturally relevant, Facebook delivered intervention to promote smoking treatment uptake and cessation among AN smokers. The Facebook content will include a digital storytelling approach adapted from the effective Centers for Disease Control (CDC) Tips from Former Smokers educational mass media campaign. The project builds on the researcher team's longstanding tobacco control research partnership with the AN community and was informed by their understanding of cultural factors that can both impede and encourage cessation in this population. If the pilot intervention is successful, researchers will have a blueprint to conduct a large randomized controlled trial. The researchers long-term objective is to develop interventions for AN tobacco users that will ultimately reduce their risk of tobacco-caused disease and mortality.

DETAILED DESCRIPTION:
The Behavioral Health Research Program at Mayo Clinic will be coordinating the study (recruit, train, oversee, etc.), but the project will take place in Alaska. The study will be conducted at the Alaska Native Tribal Health Consortium (ANTHC) in Anchorage. All data collection and the intervention will be conducted by study staff at ANTHC and Mayo Clinic. For qualitative data collection, a semi-structured interviewer guide will be developed and the project coordinator in Alaska will conduct the interviews. Researchers will provide training for the project coordinator on-site in Anchorage including 4 hours of didactic instruction followed by 4 practice hours of mock interviews and a certified completion interview. All sessions will be audiotaped. These transcripts will be coded by the researchers to assess counselor adherence to the proscribed intervention, and feedback will be provided during weekly research team teleconferences.

Mayo Clinic social media department will create the Facebook group page, develop the content library of moderator postings, and set up the software to capture participant use data. A random sample of 20% of moderator postings and responses to participant inquiries and discussions will be selected every week for the first four weeks and monthly thereafter. These transcripts will be coded by the researchers to assess moderator adherence to the proscribed intervention, and feedback will be provided during weekly research team teleconferences.

A manual of study procedures will be developed for the project coordinator in Alaska (AK). A Mayo Clinic program coordinator and clinical trials coordinator, will travel with a Mayo Clinic Co-Investigator to Anchorage, AK, to train the project coordinator on the data collection and other study procedures. The same coordination, communication, and quality control procedures will be used that have been successfully utilized in previous work. For ongoing trials in Alaska, weekly conference calls are scheduled with study staff in AK and at Mayo Clinic to discuss progress and problem solve issues related to recruitment and data collection. Quality control of the data is also monitored on site through review of participant forms and procedures every 3 months. The biostatistician on this protocol will oversee the transfer of data forms, electronic data, and data storage. The Mayo Survey Research Center will electronically transfer all data to the biostatistician. The quality of the data (data checks) including missing data and presence and frequency of outliers will be monitored once per month by the biostatistician. For study recruitment, the project coordinator will track posting of ads through Facebook (FB) and in Alaska local newsletters and websites.

All measures will be administered online using Qualtrics software, a data security service. An email link will be sent automatically by the Mayo Clinic Survey Research Center to complete the assessment. If a participant does not complete online assessments, the participant will be contacted through email or by phone by the project coordinator and prompted to complete the assessment. Data collected from survey responses will be handled and maintained by the Mayo Clinic Survey Research Center and a de-identified database of responses will be provided to the investigators. Interview forms and audio tapes will be labeled with subject ID numbers only; all personal identifiers will be removed before the data are sent to Mayo Clinic for analysis. At Mayo Clinic the audio tapes will be stored in a locked file drawer accessible only to the PI, Co-Investigator, and the project coordinator. These will be destroyed once the interviews are fully transcribed.

A trained research assistant at Mayo Clinic will mail the saliva sample kit to the participant; and the saliva samples, labeled with a subject identifier (ID) number only, will be shipped directly back to Mayo Clinic for analysis of cotinine. Once the specimen sample is processed and results posted, the sample will be destroyed immediately.

The study staff in Anchorage and Rochester will monitor any reports or observations of medical problems or severe depression or other psychiatric symptoms in participants. The Principal Investigator (PI) and a Co-Investigator from Stanford University, licensed clinical psychologists, will be consulted by telephone to consult with the study staff as needed.

ELIGIBILITY:
Inclusion and Exclusion Criteria

Participants must be:

1. >19 years of age (legal smoking age),
2. Alaska Native race/ethnicity,
3. smoke at least 1 cigarette per day over the past 7 day period,
4. if other tobacco use, cigarettes are the main tobacco product used,
5. considering or willing to make a quit attempt,
6. access to internet,
7. have an existing Facebook account or willing to set up an account, and
8. is not using pharmacotherapy or has not enrolled in a program to stop smoking for past 3 months.

   * Each person is only eligible to participate in one part of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
All data elements and data transfer activities will be strictly compliant with HIPAA privacy regulatory requirements.

REFERENCES:
- [Derived] Patten CA, Koller KR, Sinicrope PS, Prochaska JJ, Young C, Resnicow K, Decker PA, Hughes CA, Merritt ZT, McConnell CR, Huang M, Thomas TK. Facebook Intervention to Connect Alaska Native People With Resources and Support to Quit Smoking: CAN Quit Pilot Randomized Controlled Trial. Nicotine Tob Res. 2023 Mar 22;25(4):803-813. doi: 10.1093/ntr/ntac221. PMID 36130170
- [Derived] Merculieff ZT, Koller KR, Sinicrope PS, Hughes CA, Bock MJ, Decker PA, Resnicow K, Flanagan CA, Meade CD, McConnell CR, Prochaska JJ, Thomas TK, Patten CA. Developing a Social Media Intervention to Connect Alaska Native People Who Smoke with Resources and Support to Quit Smoking: The Connecting Alaska Native Quit Study. Nicotine Tob Res. 2021 May 24;23(6):1002-1009. doi: 10.1093/ntr/ntaa253. PMID 33674856
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Facebook+Quitline/Treatment Referral: * Participants join a secret/private, culturally relevant Facebook group moderated by an AN tobacco research counselor for 3 months
  * Once daily moderator postings for 30 days, repeated each month for 3 months; plus 3-4 daily check-ins/postings to respond to participant generated content and encourage sharing of personal stories/experiences relevant to all stages of the quitting process and treatment engagement
  * Description of tobacco treatment services, phone numbers and web links sent via postal mail (printed materials) and email. Treatment options provide free, professional assistance based on U.S. clinical practice guidelines: (1)AK quitline, (2)regional tribal tobacco cessation programs, and (3)smokefree.gov resources (e.g., free texting program and smartphone application, quit guide)
  Facebook Group: The pilot trial, a two-arm, parallel groups, randomized controlled design, will enroll 60 participants randomized with 1:1 allocation to the intervention or control condition. Participants will be randomized within stratified blocks based on sex (male, female), age group (19-29, 30-49, 50+ years), and region (urban, rural); potential variables related to outcomes. Assessments will be conducted for both study groups at baseline and at 1, 3, and 6 month follow-up.
Period: Overall Study
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Started | 30 | 31
Completed | 16 | 19
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.0) | 41.2 (12.9) | 40.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 30 | 31 | 61
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation Program Completion
Description: The number of participants that completed the smoking cessation program and all activities per protocol
Time Frame: 6 month follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Number analyzed (Participants) | 30 | 31
Participants | 16 | 19

2. Primary Outcome: Biochemically Confirmed Abstinence From Smoking
Description: Number of participants to have biochemically verified smoking abstinence by saliva specimen with cotinine level <15ng/ml
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Number analyzed (Participants) | 18 | 17
Participants | 2 | 2

3. Secondary Outcome: Self-reported 7-day Point Prevalence Smoking Abstinence
Description: Number of participants to self-report smoking abstinence during the past seven days (not even a puff)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Number analyzed (Participants) | 18 | 17
Participants | 7 | 3

4. Secondary Outcome: Self-reported Use of Evidence-based Cessation Treatments
Description: Number of participants to self-report use of evidence-based cessation treatments including Alaska's Tobacco Quitline, Tribal cessation programs, cessation assistance from a health care provider, nicotine replacement therapy, and other stop-smoking medications.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Number analyzed (Participants) | 18 | 17
Participants | 4 | 8

5. Secondary Outcome: Quit Attempts
Description: Number of participants to self-report a quit attempts since enrollment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
Number analyzed (Participants) | 11 | 14
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 6 months on all participants
Arm/Group | Quitline/Treatment Referral | Facebook+Quitline/Treatment Referral
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03645941/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT03645941/ICF_001.pdf